CLINICAL TRIAL: NCT03030170
Title: Does the Strengthening of the Pancreas in Distal Pancreatectomy Using Endo GIA Reload Reinforced Reduce the Occurrence of Pancreatic Fistula? Multicenter Randomized Prospective Open Study
Brief Title: REinforcement of the Pancreas in distaL pAncreatectomY (REPLAY)
Acronym: REPLAY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 35RC15_9846
Record Dates: First submitted 2017-01-16; First posted 2017-01-24 (Estimated); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Distal Pancreatectomy (DP)

STUDY DESIGN:
Intervention Model Description: intervention with reinforced medical device, or not
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Stapling of the pancreas with ENDO GIA Reinforced reload
  Interventions: Device: ENDO GIA Articulating Reinforced Reload with Tri-Staple Technology
- Control (Active Comparator): Stapling of the pancreas with ENDO GIA X-tra Thick reload
  Interventions: Device: ENDO GIA X-tra Thick reload with Tri Staple Technology

INTERVENTIONS:
Device: ENDO GIA X-tra Thick reload with Tri Staple Technology — Suture of the pancreas by normal stapling
  Arms: Control
Device: ENDO GIA Articulating Reinforced Reload with Tri-Staple Technology — Suture of the pancreas by reinforced stapling
  Arms: Experimental

SUMMARY:
Despite an improvement regarding morbidity and mortality since 30 years, especially in expert centers, pancreatic surgery remains currently associated to a significant postoperative morbidity reaching more than 60%. Regarding distal pancreatectomy (DP), the main complication following surgery is the occurrence of postoperative pancreatic fistula (PF) which may be able to lead an increased risk of bleeding, gastroparesis and finally a longer hospital stays. The main risk factors associated to the occurrence of pancreatic fistula are represented by the texture of the pancreatic parenchyma (soft pancreas) and the caliber of the main pancreatic duct (<3mm). Looking for new means of reducing the occurrence of pancreatic fistula is a priority in pancreatic surgery and a genuine public health issue. Currently, no formal recommendations concerning the optimal technical for closure of the distal stump in DP are available. In fact, manual closing by elective suturing or stapling of the main pancreatic duct give similar results. The use of a reinforcing stapling potentially represents a simple way to decrease the occurrence of pancreatic fistula and requires evaluation by a prospective randomized study.

ELIGIBILITY:
Inclusion Criteria:

* All patients who undergo DP whether made by open or laparoscopic surgery
* Patients 18 years of age or older,
* Benefiting from a social security scheme,
* Having given his free, informed and written consent.

Exclusion Criteria:

* History of pancreatic abdominal surgery
* Severe co-morbidity type renal failure requiring hemodialysis, unbalanced diabetes, major respiratory insufficiency, heart failure ≥ stage 3 NYHA;
* Persons of full age who are subject to legal protection, persons deprived of liberty.
* Pregnant or nursing women
* Patients participating in or participating in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Rate of postoperative pancreatic fistula defined by the criteria of the ISGPF | up to 90 days

SECONDARY OUTCOMES:
Gravity of the pancreatic fistula according to the 3 stages of ISGPF | up to 90 days
Assessment of the occurrence of gastroparesis and its severity according to the criteria of ISGPS | up to 90 days
Evaluation of the occurrence of postoperative haemorrhage | up to 90 days
Length of hospital stay | up to 90 days
Perioperative mortality and 90-day mortality | up to 90 days
Overall morbidity classified and categorized according to the classification of Dindo and Clavien | until 90 days
Rehospitalization rates | until 90 days

CONTACTS AND LOCATIONS:
Overall Officials: LAURENT SULPICE, MD/PHD, Principal Investigator — RENNES PONTCHAILLOU HOSPITAL
Locations (7):
- France (7):
  - Service de chirurgie Hépato-pancréato-biliaire, Clichy
  - Service de chirurgie générale, digestive et de la transplantation hépatique, Lyon
  - AP-HM - Institut Paoli Calmettes_ service de chirurgie oncologique digestive, Marseille
  - Service de chirurgie digestive et endocrienne, Nantes
  - Institut Mutualiste Montsouris, Paris
  - Centre Hospitalier Universitaire Rennes Pontchaillou, Rennes
  - Unité d'hospitalisation Chirurgie hépatique, biliaire et pancréatique, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Merdrignac A, Garnier J, Dokmak S, Regenet N, Lesurtel M, Mabrut JY, Sa Cunha A, Fuks D, Bergeat D, Robin F, Le Pabic E, Boudjema K, Turrini O, Laviolle B, Sulpice L. Effect of the Use of Reinforced Stapling on the Occurrence of Pancreatic Fistula After Distal Pancreatectomy: Results of the REPLAY (REinforcement of the Pancreas in distaL pAncreatectomY) Multicenter Randomized Clinical Trial. Ann Surg. 2022 Nov 1;276(5):769-775. doi: 10.1097/SLA.0000000000005618. Epub 2022 Jul 25. PMID 35876371